CLINICAL TRIAL: NCT01523613
Title: Clinical Performance of High-Viscous Glass-Ionomer Restorative Systems In Class II Lesions
Brief Title: High-strength Glass-ionomer Dental Restorations
Acronym: ROCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathilde Peters, DMD, PhD (Other)
Collaborators: Mott Children's Health Center (Other); Dentsply International (Industry)
Responsible Party: Sponsor-Investigator, Mathilde Peters, DMD, PhD, Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N013822; 11-PAF05343 (Other: U-Michigan)
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Dental Caries
Keywords: Dental caries; Proximal surfaces; Posterior teeth; Carious lesions; Tooth diseases; Dental restorations; Glass-ionomer
MeSH Terms: conditions — Dental Caries; Tooth Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Although material allocation was masked to evaluators, at times a difference in appearance (translucency) of the restorations at recall may have given it away.
Oversight: Data Monitoring Committee: No

ARMS (3):
- ROCK - Single Restorations (Active Comparator): ChemFil Rock glassionomer restoration
  Interventions: Device: Chemfil ROCK Glassionomer restoration
- Fuji IX GP - Single Restorations (Active Comparator): Fuji IX GP Extra glassionomer restoration
  Interventions: Device: Fuji IX GP Extra Glassionomer restoration
- Rock AND Fuji - Paired Restorations (Active Comparator): ChemFil Rock glassionomer restoration AND Fuji IX GP Extra glassionomer restoration.
  While this is not truly a separate arm for outcome analysis, this "arm" represents those individuals who had paired restorations, one of each: 1 ChemFil Rock restoration and 1 Fuji IX GP restoration.
  Interventions: Device: Chemfil ROCK Glassionomer restoration; Device: Fuji IX GP Extra Glassionomer restoration

INTERVENTIONS:
Device: Chemfil ROCK Glassionomer restoration — High-viscous glassionomer restoration of Chemfil ROCK used as posterior dental filling material.
  Other Names: HVGIC, HV-GIC, ART materials
  Arms: ROCK - Single Restorations; Rock AND Fuji - Paired Restorations
Device: Fuji IX GP Extra Glassionomer restoration — High-viscous glassionomer restoration of Fuji IX GP Extra used as posterior dental filling material.
  Other Names: Fuji Equia, HVGIC, HV-GIC, ART materials
  Arms: Fuji IX GP - Single Restorations; Rock AND Fuji - Paired Restorations

SUMMARY:
The purpose of this study is to extend our knowledge concerning the clinical performance of two dental filling materials in molars. The study will compare two high-strength glass-ionomer filling materials.

The investigators hypothesize that after two years (1) the clinical performance of both filling materials shows a similar survival rate, (2) the ChemFil Rock fillings show similar or higher incidence of fracture than Fuji IX GP fillings.

DETAILED DESCRIPTION:
In this longitudinal prospective randomized control clinical trial, posterior restorations (Class II) will be placed and evaluated for their clinical performance. The study will compare two restorative systems currently on the market in USA: both high-strength glass-ionomer (GI) restorative materials. The study restorations will be monitored for a period of up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 7-16 year old
* in need of one or two approximal fillings in molars

Exclusion Criteria:

* known allergies to calcium-aluminum-zinc-fluoro-phosphor-silicate glass or any other of glassionomer components

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde C Peters, DMD, PhD, Study Director — U Michigan
Locations (1):
- Mott Childrens' Health Center, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Restorations
Groups:
- ChemFil Rock Restoration (R): Dental restoration made of ChemFil Rock, a high-viscous glassionomer restorative used as posterior dental filling material (no cavity conditioning, no coating of finished restoration)
- Fuji IX Restoration (F): Dental restoration made of Fuji IX GP Extra, a high-viscous glassionomer restorative used as posterior dental filling material (using Cavity Conditioner and GC-Coat Plus).
- Paired Restorations (Rock + Fuji): While this is not truly a separate arm for outcome analysis, this "arm" represents those individuals who had paired restorations, one of each: 1 ChemFil Rock restorative and 1 Fuji IX GP restorative.
Period: Overall Study
Arm/Group | ChemFil Rock Restoration (R) | Fuji IX Restoration (F) | Paired Restorations (Rock + Fuji)
Started | 30; 30 Restorations (- 30 single restorations (30 R)) | 30; 30 Restorations (- 30 single restorations (30 F)) | 33; 66 Restorations (- 66 paired restorations (33R + 33F))
Completed | 23; 23 Restorations (- 23 single restorations (23R)) | 25; 25 Restorations (- 25 single restorations (25F)) | 21; 42 Restorations (- 42 paired restorations (21R and 21F))
Not Completed | 7; 7 Restorations | 5; 5 Restorations | 12; 24 Restorations

BASELINE CHARACTERISTICS:
Groups:
- ChemFil Rock Restoration (R-single): Dental restoration made of ChemFil Rock, a high-viscous glassionomer restorative used as posterior dental filling material (no cavity conditioning, no coating of finished restoration)
- Fuji IX Restoration (F-single): Dental restoration made of Fuji IX GP Extra, a high-viscous glassionomer restorative used as posterior dental filling material (using Cavity Conditioner and GC-Coat Plus).
- Paired Restorations (1R and 1F): While this is not truly a separate arm for outcome analysis, this "arm" represents those individuals who had paired restorations, one of each: 1 ChemFil Rock restorative and 1 Fuji IX GP restorative.
- Total: Total of all reporting groups
Arm/Group | ChemFil Rock Restoration (R-single) | Fuji IX Restoration (F-single) | Paired Restorations (1R and 1F) | Total
Number analyzed (Participants) | 30 | 30 | 33 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 33 | 93
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 21 | 56
  Male | 10 | 15 | 12 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 7 | 13
  Not Hispanic or Latino | 28 | 26 | 26 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 22 | 15 | 22 | 59
  White | 8 | 15 | 11 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 33 | 93

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate
Description: * Cut-off: Restoration failure as determined by (need for) replacement due to fracture and retention losses within both arms.
  * "Clinically successful" is defined as: no need for replacement due to fracture or retention losses.
Time Frame: 2 years
Population: * 21 Subjects with 2 paired restorations (21 R, 21 F).
  * 48 Subjects with a single restoration (23 R, 25 F).
  * Recall total: 69 subjects, 90 restorations.
  * No retention losses: all restorations (both R and F) in-situ and bonded; no exposed dentin.
Measure: Count of Units; unit: Restorations
Units Other Than Participants: Restorations
Groups:
- Fuji IX Restoration (F): Dental restoration made of Fuji IX GP Extra, used with Cavity Conditioner and application of GC-Coat Plus
Arm/Group | ChemFil Rock Restoration (R) | Fuji IX Restoration (F)
Number analyzed (Participants) | 44 | 46
Number analyzed (Restorations) | 44 | 46
Restorations
  Clinically successful | 39 | 44
  Replaced due to fracture | 5 | 2
  Replaced due to loss of retention | 0 | 0
Statistical Analysis 1: Comparison: ChemFil Rock Restoration (R) vs Fuji IX Restoration (F); Test type: Superiority; p = 0.262, Fisher Exact

2. Secondary Outcome: Caries Incidence Associated With Restoration
Description: - "Caries free restorations" is defined as: free of caries associated with restoration.
Time Frame: 2 years
Population: * 21 Subjects with 2 paired restorations (21 R, 21 F).
  * 48 Subjects with a single restoration (23 R, 25 F).
  * In Total: 69 subjects, 90 restorations.
Measure: Count of Units; unit: Restoration
Units Other Than Participants: Restoration
Arm/Group | ChemFil Rock Restoration (R) | Fuji IX Restoration (F)
Number analyzed (Participants) | 44 | 46
Number analyzed (Restoration) | 44 | 46
Restoration
  Caries free restorations | 40 | 39
  Restorations with caries | 4 | 7
Statistical Analysis 1: Comparison: ChemFil Rock Restoration (R) vs Fuji IX Restoration (F); Test type: Superiority; p = 0.523, Fisher Exact

3. Secondary Outcome: Restored Tooth Performance
Description: * Cut-off: Restored tooth failure (tooth in need of repair or management) as determined by Tooth integrity (enamel/tooth fracture), Sensitivity and Vitality assessment within both arms.
  * "Clinically successful" is defined as: No need for repair or management due to sensitivity or loss of tooth integrity or vitality.
Time Frame: 2 years
Population: * 21 Subjects with 2 paired restorations (21 R, 21 F).
  * 48 Subjects with a single restoration (23 R, 25 F).
Measure: Count of Units; unit: Restored tooth
Units Other Than Participants: Restored tooth
Groups:
- Rock-restored Tooth (R-tooth): Tooth restored with a ChemFil Rock filling.
- Fuji-restored Tooth (F-tooth): Tooth restored with a Fuji IX GP Extra filling.
Arm/Group | Rock-restored Tooth (R-tooth) | Fuji-restored Tooth (F-tooth)
Number analyzed (Participants) | 44 | 46
Number analyzed (Restored tooth) | 44 | 46
Restored tooth
  Clinically successful | 44 | 45
  In need of repair/management | 0 | 1
Statistical Analysis 1: Comparison: Rock-restored Tooth (R-tooth) vs Fuji-restored Tooth (F-tooth); Test type: Superiority; p = 0.100, Fisher Exact

ADVERSE EVENTS:
Time Frame: 2 years (up to 26 months in individual cases)
Groups:
- Fuji-restored (F-tooth): Tooth restored with a Fuji IX GP Extra filling.
Arm/Group | Rock-restored Tooth (R-tooth) | Fuji-restored (F-tooth)
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63

LIMITATIONS AND CAVEATS:
Current study was not designed to investigate wear behavior as final surface treatment was different between the two materials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes